CLINICAL TRIAL: NCT05896514
Title: The Role of Carotis Flow Time in Prediction of Hypotension After Anesthesia Induction in Elderly Patients
Brief Title: Carotis cFT In Prediction Of Hypotension
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, associate professor, Cukurova University
Other Study IDs: Carotid cFT
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Flow Time; Carotid Doppler Ultrasound; Hypotension; Anesthesia; Elderly
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound-guided carotid artery flow time measurement — Ultrasound-guided corrected carotid artery flow time will be measured before anestesia induction.

SUMMARY:
The aim of our study is to determine the predictive value of pre-anesthesia FTc for hypotension that may develop after general anesthesia induction in patients over 65 years of age and to investigate the correlation between pre-anesthesia FTc and the magnitude of the maximum decrease in systolic blood pressure from the pre-anaesthetic value.

DETAILED DESCRIPTION:
The FTc value of the patients to be included in the study will be measured by ultrasonography 10 minutes before the induction of anesthesia.After the measurement, the patients will be monitored with 3-lead electrocardiography, pulse oximetry and noninvasive blood pressure in the operating room. Before induction of general anesthesia, systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MAP), oxygen saturation and heart rate will measured for 3 minutes at 1-minute intervals. Induction of anesthesia with 1-2 mg/kg propofol, muscle relaxation will be achieved with 0.6 mg/kg intravenous rocuronium. During mask ventilation, 1-2% concentration of sevoflurane and 50-50% oxygen-nitrous oxide will be used. After the anesthesia induction, SBP, DBP, MAP, oxygen saturation and heart rate will be measured for 3 minutes at 1-minute intervals.

Hypotension; defined as a 30% reduction in SBP or a 20% reduction in MAP, or an absolute SBP below 90 mm Hg and MAP below 65 mm Hg within 3 minutes of induction of general anesthesia.Intravenous (iv) noradrenaline and/or iv crystalloid will be used in the treatment of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* >65 years old
* undergoing elective surgery under general anesthesia

Exclusion Criteria:

* Mean arterial pressure < 70 mmHg
* Systolic blood pressure > 180 mmHg
* Diastolic blood pressure > 110 mmHg
* < 65 years old
* Carotid artery stenosis > 50%
* ASA > 3
* Left ventricle ejection fraction < 40%
* Severe peripheral vascular disease
* Implanted pacemacer
* Autonomic nervous system disorders
* Heart valve disease
* Chronic kidney disease
* Emergency surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients > 65 years old who will undergo elective surgery under general anesthesia will be include in the study. In the preoperative unit, the FTc value in B-mode will be measured under ultrasound guidance (Esaote, MyLab tm Six Ultrasound). After the measurement, in the operating room the patients will be monitored with 3-lead electrocardiography, pulse oximetry, and noninvasive blood pressure (Infinity Kappa monitor, GE Medical Systems, Inc, Telford, PA). Before induction of anesthesia, systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MAP) and heart rate will be measured for 3 minutes at 1-minute intervals.
  Anesthesia induction will be achieved with iv 1-2 mg/kg of propofol and iv 0.6 mg/kg rocuronium will be added for muscle relaxation.Sevoflurane 1-2% and 50-50% oxygen-nitrous oxide will be used during mask ventilation. After anesthesia induction, SBP, DBP, MAP and heart rate will be measured for 3 minutes at 1-minute intervals.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
anesthesia induction related hypotension | at 1 minute after anesthesia induction, at 2 minutes after anesthesia induction, at 3 minutes anesthesia induction
  Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MAP) were measured 1 minute before anesthesia induction and after anesthesia induction (at 1 minute intervals for 3 minutes). Hypotension was defined as 30% decrease in SBP or a 20% decrease in MAP or absolute SBP less than 90 mm Hg, and MAP below 65 mm Hg within 3 minutes of induction of general anaesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)